CLINICAL TRIAL: NCT05104866
Title: A Phase-3, Open-Label, Randomized Study of Dato-DXd Versus Investigator's Choice of Chemotherapy (ICC) in Participants With Inoperable or Metastatic HR-Positive, HER2-Negative Breast Cancer Who Have Been Treated With One or Two Prior Lines of Systemic Chemotherapy (TROPION-Breast01)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9268C00001; 2023-509631-37-00 (Registry Identifier: CTIS (EU)); 2020-005620-12 (EudraCT Number)
Record Dates: First submitted 2021-10-04; First posted 2021-11-03 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; HR positive; Hormone Receptor positive; ER positive; PR positive; HER2 negative; Inoperable; Metastatic; Datopotamab Deruxtecan; Dato-DXd; DS1062; DS1062a; Capecitabine; Eribulin; Gemcitabine; Vinorelbine; TROP2; Antibody Drug Conjugate; ADC
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Capecitabine; Gemcitabine; eribulin; Vinorelbine

STUDY DESIGN:
Intervention Model Description: Parallel
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dato-DXd (Experimental): Arm 1: Dato-DXd
  Interventions: Drug: Dato-DXd
- Investigators Choice of Chemotherapy (ICC) (Active Comparator): Arm 2: ICC
  Capecitabine
  Gemcitabine
  Eribulin mesylate
  Vinorelbine
  Interventions: Drug: Capecitabine; Drug: Gemcitabine; Drug: Eribulin; Drug: Vinorelbine

INTERVENTIONS:
Drug: Dato-DXd — Experimental drug. Provided in 100mg vials. IV infusion.
  Other Names: Datopotamab deruxtecan (Dato-DXd, DS-1062a)
  Arms: Dato-DXd
Drug: Capecitabine — Tablet. Oral route of administration. Active comparator
  Arms: Investigators Choice of Chemotherapy (ICC)
Drug: Gemcitabine — IV Infusion. Active comparator
  Arms: Investigators Choice of Chemotherapy (ICC)
Drug: Eribulin — IV Infusion. Active comparator
  Other Names: Eribulin Mesylate
  Arms: Investigators Choice of Chemotherapy (ICC)
Drug: Vinorelbine — IV Infusion. Active comparator
  Arms: Investigators Choice of Chemotherapy (ICC)

SUMMARY:
The study will evaluate the safety and efficacy of datopotamab deruxtecan (also known as Dato-DXd, DS-1062a), when compared with Investigator's choice of standard of care single-agent chemotherapy (eribulin, capecitabine, vinorelbine, or gemcitabine) in participants with inoperable or metastatic HR-positive, HER2- negative breast cancer who have been treated with one or two prior lines of systemic chemotherapy.

DETAILED DESCRIPTION:
The primary objective of this study will assess the safety and efficacy of datopotamab deruxtecan (Dato-DXd) in participants with inoperable or metastatic HR-positive, HER2-negative breast cancer who have been treated with one or two prior lines of systemic chemotherapy.

The study will be stratified based on number of previous lines of chemotherapy (1 vs. 2), prior use of CDK4/6 inhibitors (Yes vs. no) and geographic region of participant (US/Canada/Europe vs. rest of world).

This study aims to see if datopotamab deruxtecan allows patients to live longer without their breast cancer getting worse, or simply to live longer, compared to patients receiving standard of care chemotherapy. This study is also looking to see how the treatment and the breast cancer affects patients' quality of life.

ELIGIBILITY:
Inclusion Criteria

Age • Participant must be ≥ 18 years at the time of screening.

Type of Participant and Disease Characteristics

* Inoperable or metastatic HR+, HER2-negative breast cancer
* Progressed on and not suitable for endocrine therapy per investigator assessment and treated with 1 to 2 lines of prior chemotherapy in the inoperable/metastatic setting. Participant must have documented progression on their most recent line of chemotherapy.
* Eligible for one of the chemotherapy options listed as ICC (eribulin, capecitabine, vinorelbine, gemcitabine), per investigator assessment.
* ECOG PS of 0 or 1, with no deterioration over the previous 2 weeks prior to day of first dosing.
* At least 1 measurable lesion not previously irradiated that qualifies as a RECIST 1.1. Note: Participants with bone-only metastases are not permitted.
* Participants with a history of previously treated neoplastic spinal cord compression, or clinically inactive brain metastases, who require no treatment with corticosteroids or anticonvulsants, may be included in the study, if they have recovered from the acute toxic effect of radiotherapy. A minimum of 2 weeks must have elapsed between the end of radiotherapy and study enrolment.
* Adequate organ and bone marrow function within 7 days before day of first dosing as follows:

  * Hemoglobin: ≥ 9.0 g/L.
  * Absolute neutrophil count: 1500/mm3.
  * Platelet count: 100000/mm3. • Total bilirubin: ≤ 1.5 × ULN if no liver metastases; or ≤ 3 × ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia) or liver metastases at baseline.
  * ALT and AST: ≤ 3 × ULN for AST/ALT; however, if elevation is due to liver metastases, ≤ 5.0 × ULN is allowed.
  * Calculated creatinine clearance: ≥ 30 mL/min as calculated using the Cockcroft-Gault equation (using actual body weight).
* LVEF ≥ 50% by either an echocardiogram or MUGA within 28 days of first dosing.
* Has had an adequate treatment washout period before Cycle 1 Day 1, defined as:

  * Major surgery: ≥ 3 weeks.
  * Radiation therapy including palliative radiation to chest: ≥ 4 weeks (palliative radiation therapy to other areas ≥ 2 weeks).
  * Anticancer therapy including hormonal therapy: ≥ 3 weeks (for small molecule targeted agents: ≥ 2 weeks or 5 half-lives, whichever is longer).
  * Antibody-based anticancer therapy: ≥ 4 weeks with the exception of receptor activator of nuclear factor kappa-B ligand (RANKL) inhibitors (eg, denosumab for the treatment of bone metastases).
  * Immunotherapy (non-antibody-based therapy): ≥ 2 weeks or 5 times the terminal elimination T½ of the agent, whichever is longer.
  * Chloroquine/hydroxychloroquine: > 14 days.
* Have available a FFPE tumor sample (block preferred, or a minimum of 20 freshly cut slides), at the time of screening. Note: Sample collection in China will comply with local regulatory approval.
* Minimum life expectancy of 12 weeks at screening.

Sex

• Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies; (oral estrogens are not permitted).

Reproduction

* Negative pregnancy test (serum) for women of childbearing potential
* Female participants must be post-menopausal for at least 1 year, surgically sterile, or using one highly effective form of birth control. Female participants must refrain from egg cell donation and breastfeeding while on study and for at least 7 months after the last dose of study intervention. Non-sterilized male partners of a woman of childbearing potential must use a male condom plus spermicide throughout this period.
* Male participants who intend to be sexually active with a female partner of childbearing potential must be surgically sterile or using a highly effective method of contraception from the time of screening throughout the total duration of the study and the drug washout period (at least 4 months after the last dose of study intervention) to prevent pregnancy in a partner. Male participants must not donate or bank sperm during this same time period. Not engaging in heterosexual activity (sexual abstinence) for the duration of the study and drug washout period is an acceptable practice if this is the preferred usual lifestyle of the participant; however, periodic or occasional abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Female partners of male participants are allowed to use HRT for contraception.

Informed Consent

* Capable of giving signed informed consent.
* Provision of signed and dated written Optional Genetic Research Information informed consent prior to collection of sample for optional genetic research that supports Genomic Initiative.

Exclusion Criteria

Medical Conditions

* Any evidence of diseases which, in the investigator's opinion, makes it undesirable for the participant to participate in the study or that would jeopardize compliance with the protocol.
* History of another primary malignancy except for malignancy treated with curative intent with no known active disease within 3 years before the first dose of study intervention and of low potential risk for recurrence. Exceptions include basal cell carcinoma of the skin and squamous cell carcinoma of the skin that has undergone potentially curative therapy, adequately resected non-melanoma skin cancer, curatively treated in situ disease, or other solid tumors curatively treated.
* Persistent toxicities caused by previous anticancer therapy (excluding alopecia), not yet improved to CTCAE Version 5.0 Grade ≤ 1 or baseline. Note: participants may be enrolled with some chronic, stable Grade 2 toxicities (defined as no worsening to > Grade 2 for at least 3 months prior to first dosing and managed with SoC treatment) which the investigator deems related to previous anticancer therapy.
* Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals; suspected infections (eg, prodromal symptoms); or inability to rule out infections.
* Known active or uncontrolled hepatitis B or C infection; or positive for hepatitis B or C virus based on the evaluation of results of tests for hepatitis B (HBsAg, anti-HBs, anti-HBc, or HBV DNA) or hepatitis C (HCV antibody or HCV RNA) infection at screening.
* Known HIV infection that is not well controlled.
* Uncontrolled or significant cardiac disease, including myocardial infarction or uncontrolled/unstable angina within 6 months prior to C1D1, CHF (New York Heart Association Class II to IV), uncontrolled or significant cardiac arrhythmia, or uncontrolled hypertension (resting systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg).
* Investigator judgment of 1 or more of the following:

  * Mean resting corrected QTcF interval > 470 ms , obtained from triplicate ECGs performed at screening.
  * History of QT prolongation associated with other medications that required discontinuation of that medication, or any current concomitant medication known to prolong the QT interval and cause Torsades de Pointes.
  * Congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives.
* History of (non-infectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder, or any autoimmune, connective tissue or inflammatory disorders with pulmonary involvement, or prior pneumonectomy.
* Leptomeningeal carcinomatosis.
* Clinically significant corneal disease.
* Known active tuberculosis infection

Prior/Concomitant Therapy

* Any of the following prior anticancer therapies:

  * Any treatment (including ADC) containing a chemotherapeutic agent targeting topoisomerase I
  * TROP2-targeted therapy
  * Prior treatment with same ICC agent
* Any concurrent anticancer treatment, with the exception of bisphosphonates, denosumab, for the treatment of bone metastases.
* Concurrent use of systemic hormonal replacement therapy (eg, estrogen). However, concurrent use of hormones for non-cancer related conditions (eg, insulin for diabetes) is acceptable.
* Major surgical procedure (excluding placement of vascular access) or significant traumatic injury within 3 weeks of the first dose of study intervention or an anticipated need for major surgery during the study.
* Receipt of live, attenuated vaccine within 30 days prior to the first dose of study treatment.

Prior/Concurrent Clinical Study Experience

* Previous treatment in the present study.
* Participation in another clinical study with a study intervention or investigational medicinal device administered in the last 4 weeks prior to first dosing, randomization into a prior Dato-DXd or T-DXd (trastuzumab deruxtecan) study regardless of treatment assignment, or concurrent enrolment in another clinical study, unless it is an observational (noninterventional) clinical study or during the follow-up period of an interventional study.
* Participants with a known hypersensitivity to Dato-DXd, or any of the excipients of the product (including, but not limited to, polysorbate 80).
* Known history of severe hypersensitivity reactions to other monoclonal antibodies.

Other Exclusions

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions and requirements.
* For women only, currently pregnant (confirmed with positive pregnancy test) or breastfeeding, or who are planning to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 732 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2026-07-31 (Estimated)

CONTACTS AND LOCATIONS:
Locations (140):
- United States (13):
  - Research Site, Duarte, California
  - Research Site, Los Angeles, California
  - Research Site, Palo Alto, California
  - Research Site, San Francisco, California
  - Research Site, Jacksonville, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Boston, Massachusetts
  - Research Site, Grand Rapids, Michigan
  - Research Site, New York, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Nashville, Tennessee
  - Research Site, Richmond, Virginia
- Argentina (5):
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, La Plata
  - Research Site, Mar del Plata
  - Research Site, Rosario
- Belgium (3):
  - Research Site, Anderlecht
  - Research Site, Leuven
  - Research Site, Liège
- Brazil (6):
  - Research Site, Itajaí
  - Research Site, Jaú
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Canada (4):
  - Research Site, North York, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- China (15):
  - Research Site, Baoding
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Jinan
  - Research Site, Linyi
  - Research Site, Nanchang
  - Research Site, Shanghai
  - Research Site, Tianjin
  - Research Site, Xiamen
- France (8):
  - Research Site, Bezannes
  - Research Site, Bordeaux
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Plérin
  - Research Site, Toulouse
  - Research Site, Villejuif
- Germany (5):
  - Research Site, Heidelberg
  - Research Site, Homburg
  - Research Site, Leipzig
  - Research Site, München
  - Research Site, Ravensburg
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Szekszárd
  - Research Site, Szolnok
- India (8):
  - Research Site, Gūrgaon
  - Research Site, Howrah
  - Research Site, Hyderabad
  - Research Site, Jaipur
  - Research Site, Kolkata
  - Research Site, Nashik
  - Research Site, Surat
  - Research Site, Visakhapatnam
- Italy (9):
  - Research Site, Bologna
  - Research Site, Candiolo
  - Research Site, Florence
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Prato
  - Research Site, Roma
- Japan (19):
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Hiroshima
  - Research Site, Isehara-shi
  - Research Site, Kagoshima
  - Research Site, Kashiwa
  - Research Site, Kitaadachi-gun
  - Research Site, Kōtoku
  - Research Site, Kyoto
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Nishinomiya-shi
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sapporo
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
  - Research Site, Yokohama
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Rotterdam
  - Research Site, Venlo
- Poland (8):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Konin
  - Research Site, Koszalin
  - Research Site, Lodz
  - Research Site, Tomaszów Mazowiecki
  - Research Site, Warsaw
- Research Site, Moscow, Russia
- South Africa (4):
  - Research Site, George
  - Research Site, Johannesburg
  - Research Site, Port Elizabeth
  - Research Site, Pretoria
- South Korea (2):
  - Research Site, Goyang-si
  - Research Site, Seoul
- Spain (9):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Bilbao (Vizcaya)
  - Research Site, Huelva
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Seville
  - Research Site, Valencia
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- United Kingdom (10):
  - Research Site, Blackpool
  - Research Site, Bristol
  - Research Site, Cardiff
  - Research Site, Colchester
  - Research Site, Edinburgh
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Nottingham
  - Research Site, Sutton
  - Research Site, Truro

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Bardia A, Jhaveri K, Im SA, Pernas S, De Laurentiis M, Wang S, Martinez Janez N, Borges G, Cescon DW, Hattori M, Lu YS, Hamilton E, Zhang Q, Tsurutani J, Kalinsky K, Rubini Liedke PE, Xu L, Fairhurst RM, Khan S, Denduluri N, Rugo HS, Xu B, Pistilli B; TROPION-Breast01 Investigators. Datopotamab Deruxtecan Versus Chemotherapy in Previously Treated Inoperable/Metastatic Hormone Receptor-Positive Human Epidermal Growth Factor Receptor 2-Negative Breast Cancer: Primary Results From TROPION-Breast01. J Clin Oncol. 2025 Jan 20;43(3):285-296. doi: 10.1200/JCO.24.00920. Epub 2024 Sep 12. PMID 39265124
- [Derived] Bardia A, Jhaveri K, Kalinsky K, Pernas S, Tsurutani J, Xu B, Hamilton E, Im SA, Nowecki Z, Sohn J, Laurentiis M, Janez NM, Adamo B, Lee KS, Jung KH, Rubovszky G, Tseng LM, Lu YS, Yuan Y, Maxwell MJ, Haddad V, Khan SS, Rugo HS, Pistilli B. TROPION-Breast01: Datopotamab deruxtecan vs chemotherapy in pre-treated inoperable or metastatic HR+/HER2- breast cancer. Future Oncol. 2024 Mar;20(8):423-436. doi: 10.2217/fon-2023-0188. Epub 2023 Jun 30. PMID 37387213
- See also: CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9268C00001&attachmentIdentifier=1ad6cc6b-d845-4b62-8243-638bb9d24742&fileName=CSP_redacted.pdf&versionIdentifier=
- See also: SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9268C00001&attachmentIdentifier=65066490-4f1f-4a60-9cc5-99164e5387da&fileName=SAP_redacted.pdf&versionIdentifier=
- See also: CSR Synopsis redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9268C00001&attachmentIdentifier=8d8f8f46-6d62-4763-8f41-e7d254349ea3&fileName=CSR_Synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Investigator's Choice of Chemotherapy (ICC): Arm 2: ICC (Capecitabine or Gemcitabine or Eribulin mesylate or Vinorelbine)
Period: Overall Study
Arm/Group | Dato-DXd | Investigator's Choice of Chemotherapy (ICC)
Started | 365 | 367
Completed | 0 | 0
Not Completed | 365 | 367
Not completed — Reason unknown | 1 | 1
Not completed — Ongoing in study at data cut-off date | 120 | 131
Not completed — Withdrawal by Subject | 25 | 29
Not completed — Lost to Follow-up | 5 | 2
Not completed — Death | 214 | 204

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dato-DXd | Investigator's Choice of Chemotherapy (ICC) | Total
Number analyzed (Participants) | 365 | 367 | 732
Age, Continuous [Median (Full Range); unit: Years] | 56.0 [29 to 86] | 54.0 [28 to 86] | 55.0 [28 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 360 | 363 | 723
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 43 | 83
  Not Hispanic or Latino | 322 | 318 | 640
  Unknown or Not Reported | 3 | 6 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    Black or African American | 4 | 7 | 11
    Native Hawaiian or other Pacific Islander | 0 | 0 | 0
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 146 | 152 | 298
    White | 180 | 170 | 350
    Other | 3 | 6 | 9
    Not reported | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: PFS is defined as time from randomization until progression per RECIST 1.1, as assessed by BICR, or death due to any cause. The analysis will include all randomized participants as randomized regardless of whether the participant withdraws from therapy, receives another anti-cancer therapy, or clinically progresses prior to RECIST 1.1.
Time Frame: On-study tumor assessments occur every 6 weeks then every 9 weeks until disease progression, death or withdrawal of consent assessed up to data cut-off (17Jul2023) to a maximum of approximately 21 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dato-DXd | Investigator's Choice of Chemotherapy (ICC)
Number analyzed (Participants) | 365 | 367
Months | 6.9 [5.7 to 7.4] | 4.9 [4.2 to 5.5]
Statistical Analysis 1: Comparison: Dato-DXd vs Investigator's Choice of Chemotherapy (ICC); Dato-DXd vs ICC; Test type: Superiority; p < 0.0001, Log Rank; Adjusted for stratification factors; Hazard Ratio (HR) = 0.63, 99% CI 2-sided [0.49 to 0.80] — Stratified Cox Proportional Hazards model. A hazard ratio < 1 favours Dato-DXd; 95% Confidence Interval 2-Sided 0.52 to 0.76

2. Primary Outcome: Overall Survival
Description: OS is defined as time from randomization until the date of death due to any cause. The comparison will include all randomized participants as randomized, regardless of whether the participant withdraws from therapy or receives another anti-cancer therapy. The measure of interest is the hazard ratio of OS.
Time Frame: From date of randomization until death due to any cause. Assessed up to data cut-off (24Jul2024) to a maximum of approximately 33 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dato-DXd | Investigator's Choice of Chemotherapy (ICC)
Number analyzed (Participants) | 365 | 367
Months | 18.6 [17.3 to 20.1] | 18.3 [17.3 to 20.5]
Statistical Analysis 1: Comparison: Dato-DXd vs Investigator's Choice of Chemotherapy (ICC); Dato-DXd vs ICC; Test type: Superiority; p = 0.9445, Log Rank — p-value adjusted for multiple testing; Adjusted for stratification factors; Hazard Ratio (HR) = 1.01, 95.97% CI 2-sided [0.83 to 1.23] — Stratified Cox Proportional Hazards model. A hazard ratio < 1 favours Dato-DXd; 95% Confidence Interval 2-Sided 0.83 to 1.22

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate is defined as the proportion of participants who have a confirmed CR or PR, as determined by the BICR/Investigator assessment, per RECIST 1.1.
Time Frame: From date of randomization until event. Assessed up to data cut-off (17Jul2023) to a maximum of approximately 21 months for BICR assessment and assessed up to data cut-off (24Jul2024) to a maximum of approximately 33 months for investigator assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Dato-DXd | Investigator's Choice of Chemotherapy (ICC)
Number analyzed (Participants) | 365 | 367
percentage of participants
  Confirmed response by BICR assessment based on IA1 data cut-off Raw Response Rate (%) | 36.44 [31.49 to 41.61] | 22.89 [18.69 to 27.53]
  Confirmed response by investigator assessment based on FA data cut-off Raw Response Rate (%) | 36.71 [31.76 to 41.89] | 22.07 [17.93 to 26.67]
Statistical Analysis 1: Comparison: Dato-DXd vs Investigator's Choice of Chemotherapy (ICC); Dato-DXd versus ICC based on confirmed response by BICR assessment based on IA1 data cut-off; Test type: Superiority; p < 0.0001, Regression, Logistic; Performed using a logistic regression model with factors for treatment and the stratification factors; Odds Ratio (OR) = 1.95, 95% CI 2-sided [1.41 to 2.71] — An odds ratio > 1 favours Dato-DXd
Statistical Analysis 2: Comparison: Dato-DXd vs Investigator's Choice of Chemotherapy (ICC); Dato-DXd versus ICC based on confirmed response by investigator assessment based on FA data cut-off; Test type: Superiority; p < 0.0001, Regression, Logistic; Performed using a logistic regression model with factors for treatment and the stratification factors; Odds Ratio (OR) = 2.06, 95% CI 2-sided [1.49 to 2.87] — An odds ratio > 1 favours Dato-DXd
Statistical Analysis 3: Comparison: Dato-DXd vs Investigator's Choice of Chemotherapy (ICC); Dato-DXd versus ICC based on confirmed response by BICR assessment based on IA1 data cut-off; Test type: Superiority; Difference in raw response rate = 13.55, 95% CI 2-sided [6.96 to 20.05] — A positive difference in response rates favours Dato-DXd. Calculated using the Miettinen-Nurminen method
Statistical Analysis 4: Comparison: Dato-DXd vs Investigator's Choice of Chemotherapy (ICC); Dato-DXd versus ICC based on confirmed response by investigator assessment based on FA data cut-off; Test type: Superiority; Difference in raw response rate = 14.64, 95% CI 2-sided [8.08 to 21.11] — A positive difference in response rates favours Dato-DXd. Calculated using the Miettinen-Nurminen method

4. Secondary Outcome: Duration of Response (DoR) as Assessed by BICR Assessment
Description: Duration of response is defined as the time from the date of first documented confirmed response until date of documented progression per RECIST 1.1, as assessed by BICR assessment or death due to any cause.
Time Frame: From date of first response until progression or death. Tumor assessments occur every 6 weeks then every 9 weeks until disease progression, death or withdrawal of consent. Assessed up to data cut-off (17Jul2023) to a maximum of approximately 21 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dato-DXd | Investigator's Choice of Chemotherapy (ICC)
Number analyzed (Participants) | 133 | 84
Months | 6.7 [5.6 to 9.8] | 5.7 [4.9 to 6.8]

5. Secondary Outcome: Duration of Response (DoR) as Assessed by Investigator Assessment
Description: Duration of response is defined as the time from the date of first documented confirmed response until date of documented progression per RECIST 1.1, as assessed by Investigator assessment or death due to any cause.
Time Frame: From date of first response until progression or death. Tumor assessments occur every 6 weeks then every 9 weeks until disease progression, death or withdrawal of consent. Assessed up to data cut-off (24Jul2024) to a maximum of approximately 33 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dato-DXd | Investigator's Choice of Chemotherapy (ICC)
Number analyzed (Participants) | 134 | 81
Months | 7.2 [5.7 to 8.6] | 6.0 [4.7 to 7.7]

6. Secondary Outcome: Progression-Free Survival by Investigator Assessment
Description: PFS by Investigator assessment will be defined as the time from the date of randomization until the date of PD per RECIST 1.1 (by Investigator assessment) or death (by any cause in the absence of progression), (ie, date of event or censoring - date of randomization + 1).
Time Frame: On-study tumor assessments occur every 6 weeks then every 9 weeks until disease progression, death or withdrawal of consent assessed up to data cut-off (24Jul2024) to a maximum of approximately 33 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dato-DXd | Investigator's Choice of Chemotherapy (ICC)
Number analyzed (Participants) | 365 | 367
Months | 6.9 [5.9 to 7.2] | 4.5 [4.2 to 5.5]
Statistical Analysis 1: Comparison: Dato-DXd vs Investigator's Choice of Chemotherapy (ICC); Dato-DXd versus ICC; Test type: Superiority; p < 0.0001, Log Rank; Adjusted for the stratification factors; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.55 to 0.76] — Stratified Cox Proportional Hazards model. A hazard ratio < 1 favours Dato-DXd

7. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants who have a confirmed CR or PR up to data cut-off date or who have SD for at least 11 weeks after randomization, per RECIST 1.1, as assessed BICR/per investigator assessment and derived from the raw tumor data.
Time Frame: Assessed up to data cut-off (17Jul2023) to a maximum of 21 months for BICR assessment and assessed up to data cut-off (24Jul2024) to a maximum of 33 months for investigator assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Dato-DXd | Investigator's Choice of Chemotherapy (ICC)
Number analyzed (Participants) | 365 | 367
percentage of participants
  Response by BICR assessment based on IA1 data cut-off Raw disease control rate (%) | 75.34 [70.59 to 79.68] | 63.76 [58.61 to 68.69]
  Response by investigator assessment based on FA data cut-off Raw disease control rate (%) | 80.82 [76.40 to 84.73] | 66.76 [61.68 to 71.56]
Statistical Analysis 1: Comparison: Dato-DXd vs Investigator's Choice of Chemotherapy (ICC); Dato-DXd versus ICC based on confirmed response by BICR assessment based on IA1 data cut-off; Test type: Superiority; p = 0.0006, Regression, Logistic; Performed using a logistic regression model with factors for treatment and the stratification factors; Odds Ratio (OR) = 1.75, 95% CI 2-sided [1.27 to 2.42] — An odds ratio > 1 favours Dato-DXd
Statistical Analysis 2: Comparison: Dato-DXd vs Investigator's Choice of Chemotherapy (ICC); Dato-DXd versus ICC based on confirmed response by Investigator assessment based on FA data cut-off; Test type: Superiority; p < 0.0001, Regression, Logistic; Performed using a logistic regression model with factors for treatment and the stratification factors; Odds Ratio (OR) = 2.12, 95% CI 2-sided [1.51 to 3.00] — An odds ratio > 1 favours Dato-DXd
Statistical Analysis 3: Comparison: Dato-DXd vs Investigator's Choice of Chemotherapy (ICC); Dato-DXd versus ICC based on confirmed response by BICR assessment based on IA1 data cut-off; Test type: Superiority; Difference in raw disease control rate = 11.58, 95% CI 2-sided [4.93 to 18.16] — A positive difference in response rates favours Dato-DXd. Calculated using the Miettinen-Nurminen method
Statistical Analysis 4: Comparison: Dato-DXd vs Investigator's Choice of Chemotherapy (ICC); Dato-DXd versus ICC based on confirmed response by Investigator assessment based on FA data cut-off; Test type: Superiority; Difference in raw disease control rate = 14.06, 95% CI 2-sided [7.74 to 20.33] — A positive difference in response rates favours Dato-DXd. Calculated using the Miettinen-Nurminen method

8. Secondary Outcome: Time to First Subsequent Therapy (TFST)
Description: Time to first subsequent therapy is defined as the time from randomization until the start date of the first subsequent anti-cancer therapy after discontinuation of randomized treatment, or death due to any cause.
Time Frame: From randomization to start of first subsequent anti-cancer therapy. Assessments occur at every visit after study treatment has been discontinued. Assessed up to data cut-off (24Jul2024) to a maximum of approximately 33 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dato-DXd | Investigator's Choice of Chemotherapy (ICC)
Number analyzed (Participants) | 365 | 367
Months | 8.0 [7.2 to 8.8] | 5.2 [4.6 to 5.8]
Statistical Analysis 1: Comparison: Dato-DXd vs Investigator's Choice of Chemotherapy (ICC); Dato-DXd versus ICC; Test type: Superiority; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.50 to 0.68] — Stratified Cox Proportional Hazards model. A hazard ratio < 1 favours Dato-DXd

9. Secondary Outcome: Time to Second Subsequent Therapy (TSST)
Description: Time to second subsequent therapy is defined as the time from randomization to until the start date of the second subsequent anti-cancer therapy after discontinuation of first subsequent treatment, or death due to any cause.
Time Frame: From randomization to start of second subsequent anti-cancer therapy. Assessments occur at every visit after study treatment has been discontinued. Assessed up to data cut-off (24Jul2024) to a maximum of approximately 33 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dato-DXd | Investigator's Choice of Chemotherapy (ICC)
Number analyzed (Participants) | 365 | 367
Months | 13.7 [12.4 to 15.0] | 12.3 [10.8 to 13.7]
Statistical Analysis 1: Comparison: Dato-DXd vs Investigator's Choice of Chemotherapy (ICC); Dato-DXd versus ICC; Test type: Superiority; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.70 to 0.98] — Stratified Cox Proportional Hazards model. A hazard ratio < 1 favours Dato-DXd

10. Secondary Outcome: Time From Randomization to Second Progression or Death (PFS2)
Description: Time to second progression of death will be defined as the time from the randomization to the earliest of the progression event (following the initial progression), subsequent to first subsequent therapy, or death. The date of second progression will be recorded by the Investigator in the eCRF and defined according to local standard clinical practice.
Time Frame: From date of randomization to second progression or death. PFS2 assessments occur every 3 months after disease progression. Assessed up to data cut-off (24Jul2024) to a maximum of approximately 33 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dato-DXd | Investigator's Choice of Chemotherapy (ICC)
Number analyzed (Participants) | 365 | 367
Months | 11.7 [10.8 to 13.1] | 10.4 [9.6 to 11.5]
Statistical Analysis 1: Comparison: Dato-DXd vs Investigator's Choice of Chemotherapy (ICC); Dato-DXd versus ICC; Test type: Superiority; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.63 to 0.93] — Stratified Cox Proportional Hazards model. A hazard ratio < 1 favours Dato-DXd

11. Secondary Outcome: Clinical Outcome Assessment- TTD in Pain
Description: Time to deterioration in pain as measured by the pain scale from EORTC QLQ-C30. Deterioration is defined as a 16.6 increase in score relative to baseline score
Time Frame: From date of randomization to 18 weeks post-progression. Assessments occur every 3 weeks then every 6 weeks until 18 weeks post-progression and at end of treatment visit. Assessed up to data cut-off (24Jul2024) to a maximum of approximately 33 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dato-DXd | Investigator's Choice of Chemotherapy (ICC)
Number analyzed (Participants) | 365 | 367
Months | 3.5 [2.8 to 5.0] | 2.8 [2.1 to 3.4]
Statistical Analysis 1: Comparison: Dato-DXd vs Investigator's Choice of Chemotherapy (ICC); Dato-DXd versus ICC; Test type: Superiority; p = 0.1519, Log Rank; Adjusted for stratification factors; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.67 to 1.06] — Stratified Cox Proportional Hazards model. A hazard ratio < 1 favours Dato-DXd

12. Secondary Outcome: Clinical Outcome Assessment- TTD in Physical Functioning
Description: Time to deterioration in physical functioning as measured by the physical functioning scale from EORTC QLQ-C30. Deterioration is defined as a 13.3 decrease in score relative to baseline score.
Time Frame: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dato-DXd | Investigator's Choice of Chemotherapy (ICC)
Number analyzed (Participants) | 365 | 367
Months | 5.6 [3.5 to 9.7] | 3.5 [2.2 to 4.9]
Statistical Analysis 1: Comparison: Dato-DXd vs Investigator's Choice of Chemotherapy (ICC); Dato-DXd versus ICC; Test type: Superiority; p = 0.0596, Log Rank; Adjusted for stratification factors; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.62 to 1.01] — Stratified Cox Proportional Hazards model. A hazard ratio < 1 favours Dato-DXd

13. Secondary Outcome: Clinical Outcome Assessment- TTD in GHS
Description: Time to deterioration in global health status/QoL as measured by the global health status/QoL scale from EORTC QLQ-C30. Deterioration is defined as a 16.6 decrease in score relative to baseline score.
Time Frame: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dato-DXd | Investigator's Choice of Chemotherapy (ICC)
Number analyzed (Participants) | 365 | 367
Months | 3.4 [2.1 to 5.0] | 2.1 [1.5 to 2.9]
Statistical Analysis 1: Comparison: Dato-DXd vs Investigator's Choice of Chemotherapy (ICC); Dato-DXd versus ICC; Test type: Superiority; p = 0.1155, Log Rank; Adjusted for stratification factors; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.67 to 1.04] — Stratified Cox Proportional Hazards model. A hazard ratio < 1 favours Dato-DXd

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected from time of signature of informed consent until the follow-up period is completed (35 days after the last dose of study treatment) (maximum duration of approximately 28 months). All-Cause Mortality was assessed up to data cut-off (24Jul2024) to a maximum of approximately 33 months.
Description: All-Cause Mortality was assessed in the Full Analysis Set (all randomised participants). Serious and Other adverse events were assessed in the Safety Analysis Population (all treated subjects)
Arm/Group | Dato-DXd | Investigator's Choice of Chemotherapy (ICC)
All-Cause Mortality (participants affected / at risk) | 223/365 | 213/367
Serious Adverse Events (participants affected / at risk) | 62/360 | 67/351
Other Adverse Events (participants affected / at risk) | 348/360 | 329/351
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dato-DXd (N=360) | Investigator's Choice of Chemotherapy (ICC) (N=351)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 1 (1)
Hypercalcaemia of malignancy (Endocrine disorders) | 0 (0) | 1 (1)
Thyroiditis subacute (Endocrine disorders) | 1 (2) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Punctate keratitis (Eye disorders) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastric mucosal lesion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip blister (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder rupture (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 4 (4) | 3 (3)
Covid-19 pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Coronavirus pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (2)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (3) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Meningitis tuberculous (Infections and infestations) | 0 (0) | 1 (1)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 4 (4)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 2 (2)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 2 (2)
Spinal cord infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (7) | 3 (4)
Urosepsis (Infections and infestations) | 3 (4) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Radiation necrosis (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes with hyperosmolarity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dato-DXd (N=360) | Investigator's Choice of Chemotherapy (ICC) (N=351)
Dysgeusia (Nervous system disorders) | 19 (21) | 14 (14)
Headache (Nervous system disorders) | 30 (35) | 38 (46)
Neuropathy peripheral (Nervous system disorders) | 6 (6) | 24 (28)
Paraesthesia (Nervous system disorders) | 10 (10) | 21 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 49 (58) | 33 (36)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 22 (23)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 22 (36) | 6 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 136 (139) | 80 (80)
Dry skin (Skin and subcutaneous tissue disorders) | 23 (23) | 6 (6)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 9 (9) | 45 (52)
Pruritus (Skin and subcutaneous tissue disorders) | 32 (37) | 7 (8)
Rash (Skin and subcutaneous tissue disorders) | 34 (35) | 10 (11)
Blepharitis (Eye disorders) | 28 (28) | 6 (7)
Dry eye (Eye disorders) | 97 (107) | 46 (47)
Keratitis (Eye disorders) | 30 (37) | 10 (15)
Lacrimation increased (Eye disorders) | 28 (29) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 62 (78) | 86 (134)
Meibomian gland dysfunction (Eye disorders) | 25 (27) | 6 (6)
Punctate keratitis (Eye disorders) | 43 (53) | 23 (26)
Abdominal pain (Gastrointestinal disorders) | 25 (28) | 30 (33)
Constipation (Gastrointestinal disorders) | 126 (161) | 60 (70)
Diarrhoea (Gastrointestinal disorders) | 41 (59) | 67 (95)
Dry mouth (Gastrointestinal disorders) | 21 (32) | 6 (6)
Nausea (Gastrointestinal disorders) | 204 (326) | 95 (126)
Stomatitis (Gastrointestinal disorders) | 188 (300) | 49 (58)
Vomiting (Gastrointestinal disorders) | 86 (118) | 41 (59)
Asthenia (General disorders) | 56 (97) | 61 (72)
Fatigue (General disorders) | 102 (117) | 71 (80)
Pyrexia (General disorders) | 29 (33) | 38 (52)
Leukopenia (Blood and lymphatic system disorders) | 13 (25) | 29 (61)
Covid-19 (Infections and infestations) | 70 (75) | 50 (51)
Upper respiratory tract infection (Infections and infestations) | 21 (25) | 19 (20)
Urinary tract infection (Infections and infestations) | 24 (31) | 18 (20)
Neutropenia (Blood and lymphatic system disorders) | 21 (29) | 91 (194)
Alanine aminotransferase increased (Investigations) | 38 (50) | 50 (68)
Aspartate aminotransferase increased (Investigations) | 61 (78) | 59 (80)
Blood alkaline phosphatase increased (Investigations) | 22 (28) | 16 (24)
Neutrophil count decreased (Investigations) | 25 (58) | 75 (205)
Platelet count decreased (Investigations) | 9 (11) | 18 (28)
Weight decreased (Investigations) | 31 (32) | 16 (17)
White blood cell count decreased (Investigations) | 18 (37) | 41 (114)
Decreased appetite (Metabolism and nutrition disorders) | 58 (77) | 55 (64)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (24) | 25 (28)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 22 (23)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 23 (25)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 (24) | 21 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-04-22): https://cdn.clinicaltrials.gov/large-docs/66/NCT05104866/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-17): https://cdn.clinicaltrials.gov/large-docs/66/NCT05104866/SAP_001.pdf